CLINICAL TRIAL: NCT04646291
Title: Retrospective Study on the Use, Efficiency, and Safety of the At-home Mosie Kit
Status: Completed | Type: Observational
Sponsor: Mosie Baby (Industry)
Responsible Party: Principal Investigator, Karina Loyo PhD MBA CCDM, Research Consultant, Mosie Baby
Other Study IDs: Mosie-001
Record Dates: First submitted 2020-08-13; First posted 2020-11-27 (Actual); Results first posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Infertility; Infertility, Female; Infertility, Male
Keywords: Insemination; Infertility; Pregnancy
MeSH Terms: conditions — Infertility; Infertility, Female; Infertility, Male

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Heterosexual Females with a Male partner: This cohort consists of heterosexual females with a male partner who have used the Mosie Baby Kit for insemination during at least one cycle
  Interventions: Device: Insemination with the Mosie Baby Kit
- Females in LGBTQ Relationships: This cohort consists of females in LGBTQ Relationships who have used the Mosie Baby Kit for insemination during at least one cycle.
  Interventions: Device: Insemination with the Mosie Baby Kit
- Solo parent: This generally will be a female without a partner who has used the Mosie Baby Kit for insemination during at least one cycle. However, it might also be a male who is using a surrogate female.
  Interventions: Device: Insemination with the Mosie Baby Kit

INTERVENTIONS:
Device: Insemination with the Mosie Baby Kit — The participant will have performed at least one cycle of insemination using the Mosie Baby Kit.

SUMMARY:
This study examines the experience of people who have selected to use the at-home insemination Mosie Kit to understand the user's experience, the perceived safety and the efficiency. People who have recently purchased and voluntarily selected to use the Mosie Kit will be invited to complete a one-time online anonymous survey. The results of the survey will be analyzed to understand their experiences.

DETAILED DESCRIPTION:
At-home intracervical insemination (ICI), folklorickly known as the "turkey-baster" method, has been used for decades to increase likelihood of pregnancy. This method works by depositing semen close to or at the cervix. While there are several devices such as over the counter syringes and silicone caps, the creator of the Mosie Baby syringe believes it is designed to be more ergonomic and compatible with a woman's body, easy and safe to use, and results in depositing the semen at or near the cervix opening. The Mosie Kit provides people with an at-home intracervical insemination option which could be used before resorting to more invasive and expensive options such as Intrauterine Insemination (IUI) or in vitro fertilization. There is vast evidence of Mosie's success in the form of happy users who have conceived. There is a desire to learn more about the safety, useability and experience of using the Mosie kit.

This retrospective study will examine the experience of people who have voluntarily chosen to purchase and use the Mosie Kit. The Mosie Kit consists of 2 syringes and a semen collection cup Understanding the safety, useability and experience of using the Mosie Kit will provide additional information about the nature of using intracervical insemination as a viable method for getting pregnant. The information gained will increase understanding of how viable the Mosie Kit is as a first step in trying to conceive and how it is perceived by the people who have chosen to use it.

ELIGIBILITY:
Inclusion Criteria:

* Provide implicit consent by filling out and submitting the survey.
* Used a Mosie Kit to conceive during at least one cycle.
* At least 18 years old.
* Has an active email on file (presumed or they would not have received an invitation to participate. This information will not be verified as there is a desire to keep the survey completely anonymous.)

Exclusion Criteria:

* Never used a Mosie Kit

Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of all individuals who have purchased the Mosie Kit in the past 2-8 complete months prior to study initiation. All qualifying individuals will receive an invitation to participate. These individuals will typically be of child-bearing age, both females and males, and generally ages ranging 18-50 years old.
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karina Loyo, PhD MBA CCDM, Principal Investigator — Independent Researcher
Locations (1):
- Virtual Study - Online Data Collection, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Currently there is no plan to share data.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A retrospective study of people who had purchased the Mosie Kit between October 2019 and July 2020 was conducted to understand the efficacy, safety and usability of the at-home insemination kit. Participants were recruited in August 2020 via emailed invitation.
Pre-assignment Details: Subjects who were 18 years old and who had used the at-home Mosie Insemination kit for at least one cycle were included in the study.
Period: Overall Study
Arm/Group | Heterosexual Females With a Male Partner | Females in LGBTQ Relationships | Solo Parent
Started | 272 | 70 | 8
Completed | 272 | 70 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Heterosexual Females With a Male Partner: This cohort consists of heterosexual females with a male partner who have used the Mosie Baby Kit for insemination during at least one cycle Insemination with the Mosie Baby Kit: The participant will have performed at least one cycle of insemination using the Mosie Baby Kit.
- Total: Total of all reporting groups
Arm/Group | Heterosexual Females With a Male Partner | Females in LGBTQ Relationships | Solo Parent | Total
Number analyzed (Participants) | 272 | 70 | 8 | 350
Age, Customized [Count of Participants; unit: Participants]
  20-24 years old | 6 | 5 | 0 | 11
  25-29 years old | 39 | 20 | 1 | 60
  30-34 years old | 83 | 30 | 2 | 115
  35-39 years old | 100 | 10 | 3 | 113
  40-45 years old | 41 | 5 | 1 | 47
  45-50 years old | 4 | 0 | 0 | 4
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 255 | 65 | 8 | 328
  Male | 17 | 0 | 0 | 17
  Non-binary (female) | 0 | 2 | 0 | 2
  Transgender (female) | 0 | 2 | 0 | 2
  Transgender (male) | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Participants were allowed to select all that applied from the options which include the categories listed plus Hispanic/LatinX. The other category below reports those that selected only Hispanic/LatinX plus other as a category. The Multiple Race reflects all that selected either multiple race or more than one race or ethnicity.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 14 | 0 | 0 | 14
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 25 | 11 | 0 | 36
    White | 178 | 35 | 5 | 218
    More than one race | 16 | 14 | 2 | 32
    Unknown or Not Reported | 39 | 10 | 1 | 50
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 272 | 70 | 8 | 350
Cycles Analyzed [Count of Participants; unit: Participants]
  1 Cycle | 98 | 39 | 4 | 141
  2 cycles | 88 | 14 | 2 | 104
  3 cycles | 53 | 8 | 0 | 61
  4 cycles | 16 | 4 | 0 | 20
  5 cycles | 13 | 3 | 0 | 16
  6 cycles | 4 | 2 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Pregnancy Rate
Description: The study will measure whether using the Mosie Baby Kit for insemination will result in pregnancy.
Time Frame: Up to 6 full menstrual cycles (generally 28 days in length) prior to survey. The number of cycles reported by each participant may vary.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: The retrospective study examined 350 qualified participants. Females and males, non-binary, and transgender people were included in the study. The information provided includes all 3 arms unless specified.
Arm/Group | All Participants | Heterosexual Females With a Male Partner | Females in LGBTQ Relationships | Solo Parent
Number analyzed (Participants) | 350 | 272 | 70 | 8
Participants
  Number of Participants Achieving Pregnancy | 99 | 71 | 24 | 4
  Number of Participants Not Getting Pregnant | 251 | 201 | 46 | 4

2. Primary Outcome: Cycle in Which Pregnancy Was Reported
Description: The outcome measure is the number of cycles of Mosie use which resulted in a positive pregnancy test.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Pregnancies: This subgroup represents the women who ended up pregnant as a result of using Mosie.
Arm/Group | Pregnancies | Heterosexual Females With a Male Partner | Females in LGBTQ Relationships | Solo Parent
Number analyzed (Participants) | 99 | 71 | 24 | 4
Participants
  1 cycle resulted in a pregnancy | 60 | 46 | 12 | 2
  2 cycles resulted in a pregnancy | 18 | 12 | 5 | 1
  3 cycles resulted in a pregnancy | 13 | 9 | 4 | 0
  4 cycles resulted in a pregnancy | 1 | 1 | 0 | 0
  5 cycles resulted in a pregnancy | 0 | 0 | 0 | 0
  6 cycles resulted in a pregnancy | 4 | 2 | 1 | 1
  6+ cycles resulted in a pregnancy | 3 | 1 | 2 | 0

3. Primary Outcome: Pregnancy Rate Differences Between Couples With Fertility Issues and Without
Description: The study will measure the difference in pregnancy rates of Mosie Baby Kit users with known fertility issues and those without known fertility issues.
Time Frame: as for outcome 1
Population: The number differs because the denominator shows the number of women fitting each of the described criteria. This adjustment is required in order to be able to examine this hypothesis which is based on the rate of each group's pregnancy rate.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants | Heterosexual Females With a Male Partner | Females in LGBTQ Relationships | Solo Parent
Number analyzed (Participants) | 350 | 272 | 70 | 8
Participants
  Participants with no fertility issue who got pregnant | 69 | 44 | 21 | 4
  Participants with no fertility issue who did not get pregnant | 134 | 89 | 42 | 3
  Participants with a fertility issues who got pregnant | 31 | 27 | 3 | 1
  Participants with a fertility issues who did not get pregnant | 116 | 112 | 4 | 0

4. Secondary Outcome: Ease of Use
Description: The study will examine the perceived ease of use of the Mosie Kit.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants | Heterosexual Females With a Male Partner | Females in LGBTQ Relationships | Solo Parent
Number analyzed (Participants) | 350 | 272 | 70 | 8
Participants
  Easy Process Overall: Strongly Disagree | 0 | 0 | 0 | 0
  Easy Process Overall: Disagree | 2 | 0 | 2 | 0
  Easy Process Overall: Neutral | 7 | 6 | 1 | 0
  Easy Process Overall: Agree | 101 | 85 | 14 | 2
  Easy Process Overall: Strongly Agree | 240 | 181 | 53 | 6
  Intuitive Process: Strongly Disagree | 0 | 0 | 0 | 0
  Intuitive Process: Disagree | 13 | 10 | 3 | 0
  Intuitive Process: Neutral | 19 | 18 | 0 | 1
  Intuitive Process: Agree | 121 | 100 | 18 | 3
  Intuitive Process: Strongly Agree | 197 | 144 | 49 | 4

5. Secondary Outcome: Ease of Use: Usage Steps
Description: The use of the Mosie Kit requires several steps. In order to examine ease of use, each step was also examined individually. This table reports the data associated with each of use during each step of the insemination process.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants | Heterosexual Females With a Male Partner | Females in LGBTQ Relationships | Solo Parent
Number analyzed (Participants) | 350 | 272 | 70 | 8
Participants
  Easy Sample Collection: Very Difficult | 3 | 1 | 2 | 0
  Easy Sample Collection: Difficult | 16 | 15 | 1 | 0
  Easy Sample Collection: Neutral | 32 | 18 | 11 | 3
  Easy Sample Collection: Easy | 112 | 90 | 21 | 1
  Easy Sample Collection: Very Easy | 187 | 148 | 35 | 4
  Draw up Semen: Very Difficult | 2 | 0 | 2 | 0
  Draw up Semen: Difficult | 7 | 3 | 4 | 0
  Draw up Semen: Neutral | 31 | 23 | 7 | 1
  Draw up Semen: Easy | 128 | 104 | 23 | 1
  Draw up Semen: Very Easy | 182 | 142 | 34 | 6
  Insert Syringe: Very Difficult | 0 | 0 | 0 | 0
  Insert Syringe: Difficult | 2 | 1 | 1 | 0
  Insert Syringe: Neutral | 8 | 7 | 0 | 1
  Insert Syringe: Easy | 108 | 91 | 16 | 1
  Insert Syringe: Very Easy | 232 | 173 | 53 | 6
  Deposit Sperm: Very Difficult | 0 | 0 | 0 | 0
  Deposit Sperm: Difficult | 10 | 7 | 3 | 0
  Deposit Sperm: Neutral | 24 | 20 | 3 | 1
  Deposit Sperm: Easy | 105 | 87 | 17 | 1
  Deposit Sperm: Very Easy | 211 | 158 | 47 | 6

6. Secondary Outcome: Use of the Kit as Intended
Description: The study will examine whether the user's used the Mosie Kit as described in the instructions and as intended.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: The retrospective study examined 350 qualified participants. Females and males, non-binary, and transgender people were included in the study. The information provided includes all 3 arms.
Arm/Group | All Participants | Heterosexual Females With a Male Partner | Females in LGBTQ Relationships | Solo Parent
Number analyzed (Participants) | 350 | 272 | 70 | 8
Participants
  Read instructions | 333 | 258 | 67 | 8
  Prepared items | 333 | 256 | 69 | 8
  Washed my hands | 324 | 251 | 65 | 8
  Tested syringe | 305 | 234 | 63 | 8
  Partner washed hands | 288 | 225 | 59 | 4

7. Secondary Outcome: Perceived Safety of Using the Mosie Kit
Description: The study will examine the user's perceived safety of using the Mosie Kit syringe by evaluating overall perceived safety.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants | Heterosexual Females With a Male Partner | Females in LGBTQ Relationships | Solo Parent
Number analyzed (Participants) | 350 | 272 | 70 | 8
Participants
  Strongly Disgree | 0 | 0 | 0 | 0
  Disagree | 1 | 1 | 0 | 0
  Neutral | 2 | 2 | 0 | 0
  Agree | 95 | 80 | 13 | 2
  Strongly Agree | 252 | 189 | 57 | 6

8. Other Pre Specified Outcome: Pregnancy Rate Comparison Between Male Infertility Source and Female Infertility Source or Unknown Infertility Status
Description: The study will examine the resulting pregnancy rates of users self-identified as having a male infertility issue versus those having a female infertility issue and those having no reported fertility issue.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- All Pregnant Participants: Reflects only the pregnant participants
Arm/Group | All Pregnant Participants | Heterosexual Females With a Male Partner | Females in LGBTQ Relationships | Solo Parent
Number analyzed (Participants) | 99 | 71 | 24 | 4
Participants
  Pregnancies to participants with Issues of Female Origin | 25 | 20 | 3 | 2
  Pregnancies to participants with Issues of Male origin | 11 | 8 | 3 | 0
  Pregnancies to participants No infertility Issue | 59 | 39 | 18 | 2
  Pregnancies to participantsBoth Male and Female Infertility Issue | 4 | 4 | 0 | 0

9. Other Pre Specified Outcome: Comparison of Pregnancy Rate Based on Known Fertility Issue
Description: The study will examine the resulting pregnancy rates of users in comparison to the type of infertility issue reported.
Time Frame: as for outcome 1
Population: All participants reporting a pregnancy were asked to indicate as many sources of infertility as desired by marking the options provided. Some participants reported multiple sources for their fertility issue (n=48). Also some participants noted 'No' fertility issue (n=51). The outcome data table shows all conditions available for selection plus a row to capture the participants that indicated no infertility source. Data can only be aggregated across a row; data should not be aggregated by column.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants | Heterosexual Females With a Male Partner | Females in LGBTQ Relationships | Solo Parent
Number analyzed (Participants) | 99 | 71 | 24 | 4
Participants
  PCOS | 12 | 8 | 3 | 1
  Endometriosis Low AMH or low ovarian reserve | 4 | 4 | 0 | 0
  Vaginismus or vulvodynia | 6 | 6 | 0 | 0
  Tilted Uterus | 4 | 4 | 0 | 0
  Low Sperm Count | 6 | 5 | 1 | 0
  Sperm motility issues | 4 | 4 | 0 | 0
  Erectile Dysfunction | 5 | 5 | 0 | 0
  Performance issues or sexual anxiety, or inability to orgasm with partner | 14 | 14 | 0 | 0
  Unexplained infertility | 10 | 9 | 0 | 0
  No fertility issues reported | 51 | 32 | 17 | 2

10. Other Pre Specified Outcome: Insemination Schedule's Impact on Pregnancy
Description: The study examined pregnancy rates of users inseminating twice as expected as compared to using a different schedule. Four time points within each cycle were examined: 24-48 hours before ovulation, within 24 hours of ovulation, 24-48 hours after ovulation and 48 or more hours after ovulation. The recommended time frame is at least 2 insemination during the aggregate of 24-48 hours prior to ovulation and the within 24 hours of ovulation. The table below shows the data for how many women met the insemination criteria for each cycle that reported being pregnant.
  Note: Number of cycles reported by women vary from 1 cycle to 6 cycles. it is possible that a participant may have met the criteria at one cycle and not the other. Given this, the 3 arms when aggregated per row will equal the total of all participants. However, columns will not add up to the total participants per arm.
Time Frame: as for outcome 1
Population: Only participants who ended up pregnant are included in this analysis.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: The retrospective study examined 350 qualified participants. Females and males, non-binary, and transgender people were included in the study.
Arm/Group | All Participants | Heterosexual Females With a Male Partner | Females in LGBTQ Relationships | Solo Parent
Number analyzed (Participants) | 99 | 71 | 24 | 4
Participants
  1st cycle : at least 2 inseminations per cycle | 52 | 30 | 10 | 2
  1st cycle not meeting criteria | 47 | 41 | 14 | 2
  1st cycle not reporting | 0 | 0 | 0 | 0
  2nd cycles : at least 2 inseminations per cycle | 18 | 13 | 4 | 1
  2nd cycle not meeting criteria | 24 | 16 | 6 | 2
  2nd cycle not reporting | 57 | 42 | 14 | 1
  3rd cycles : at least 2 inseminations per cycle | 5 | 4 | 1 | 0
  3rd cycle not reporting | 83 | 62 | 18 | 3
  3rd cycle not meeting criteria | 11 | 5 | 5 | 1
  4th cycles : at least 2 inseminations per cycle | 4 | 4 | 0 | 0
  4th cycle not meeting criteria | 2 | 1 | 0 | 1
  4th cycle not reporting | 93 | 66 | 24 | 3
  5th cycles : at least 2 inseminations per cycle | 0 | 0 | 0 | 0
  5th cycle not meeting criteria | 0 | 0 | 0 | 0
  5th cycle not reporting | 99 | 71 | 24 | 4
  6th cycles : at least 2 inseminations per cycle | 1 | 0 | 0 | 1
  6th cycle not meeting criteria | 0 | 0 | 0 | 0
  6th cycle not reporting | 98 | 71 | 24 | 3

11. Other Pre Specified Outcome: Effect of COVID on Family Expansion
Description: The study will examine the effect of COVID on family expansion plans. The analysis will be provided in aggregate because the focus is on the impact of COVID on family expansion overall and not on whether one arm has more or less impact. This is a tertiary exploratory measure that does not evaluate the core product.
Time Frame: Pregnancies reported as conceived using the Mosie Kit during the months of December 2019 to February 2020 (Pre-COVID) will be compared to those reported for March - July 2020 (during COVID).
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: The retrospective study examined 350 qualified participants. Females and males, non-binary, and transgender people were included in the study. The information provided includes all 3 arms because the focus of this questions is on the impact of COVID without regard for sexual preference.
Arm/Group | All Participants | Heterosexual Females With a Male Partner | Females in LGBTQ Relationships | Solo Parent
Number analyzed (Participants) | 350 | 272 | 70 | 80
Participants
  Yes | 89 | 67 | 22 | 0
  No | 261 | 205 | 48 | 8

12. Other Pre Specified Outcome: Pregnancy Outcomes During COVID
Description: The study will examine whether there were more or less pregnancy rates during COVID. This measure will be an aggregate measure of all women. It is an exploratory measure to understand the impact of COVID. No data will be provided by study arm.
Time Frame: Pregnancies reported as conceived using the Mosie Kit during the months of September 2019 to February 2020 (Pre-COVID) will be compared to those reported for March - August 2020 (during COVID).
Measure: Count of Participants; unit: Participants
Groups:
- Pregnancies: This subgroup represents the women who ended up pregnant as a result of using Mosie. The information provided includes all women from all 3 arms because the focus of this questions is on the impact of COVID without regard for sexual preference.
Arm/Group | Pregnancies | Heterosexual Females With a Male Partner | Females in LGBTQ Relationships | Solo Parent
Number analyzed (Participants) | 99 | 71 | 24 | 8
Participants
  Conception: September 2019 Birth: June 2020 | 1 | 0 | 1 | 0
  Conception: October 2019 Birth: July 2020 | 3 | 2 | 1 | 0
  Conception: November 2019 Birth: August 2020 | 5 | 2 | 3 | 0
  Conception: December 2019 Birth: August 2020 | 4 | 3 | 0 | 1
  Conception: January 2020 Birth: September 2021 | 3 | 2 | 1 | 0
  Conception: February 2020 Birth: November 2021 | 10 | 5 | 5 | 0
  Conception: March 2020 Birth: December 2021 | 7 | 5 | 2 | 0
  Conception: April 2020 Birth: Jan 2021 | 16 | 12 | 2 | 2
  Conception: May 2020 Birth: Feb 2021 | 11 | 8 | 3 | 0
  Conception: June 2020 Birth: March 2021 | 19 | 14 | 5 | 0
  Conception: July 2020 Birth: April 2021 | 17 | 15 | 1 | 1
  Conception: August 2020 Birth: May 2021 | 2 | 2 | 0 | 0
  Unknown | 1 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: No adverse events were reported specifically for this retrospective study.
Description: Adverse events were not collected for this retrospective study. All-cause mortality was not collected and is not recorded for this study.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-07-31): https://cdn.clinicaltrials.gov/large-docs/91/NCT04646291/Prot_SAP_ICF_000.pdf